CLINICAL TRIAL: NCT04810663
Title: Outcome of Radiation Therapy In Operated Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ezzat Mohamed, principal Investigator, Assiut University
Other Study IDs: Radiotherapy in gastric cancer
Record Dates: First submitted 2021-03-08; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Adjuvant Radiotherapy in operated gastric cancer

SUMMARY:
* Study tolerability and toxicity of radiotherapy with or without chemotherapy for operated gastric cancer.
* Evaluate the efficacy of adjuvant radiotherapy with or without chemotherapy as regarding local control and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient; ≥18 and ≤75 years.
* Histologically proven gastric or gastroesophageal adenocarcinoma.
* Pt received adjuvant Radiotherapy with or without chemotherapy with any protocol.

Exclusion Criteria:

* Patient >75 years&<18 years.
* Histologically types other than adenocarcinoma .
* Metastatic patients (M1).
* Pt didn't recive radiotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age of the patient; ≥18 and ≤75 years. Histologically proven gastric or gastroesophageal adenocarcinoma. Pt received adjuvant Radiotherapy with or without chemotherapy with any protocol.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Radiotherapy in operated gastric cancer | Baseline
  Disease Free Survival

REFERENCES:
- [Result] 1- A. Schernberg,a E. Rivin del Campo,a B. Rousseau,b O. Matzinger,c M. Loi,d P. Maingon,e,f and F. Hugue. Adjuvant chemoradiation for gastric carcinoma: State of the art and perspectives. ClinTranslRadiatOncol. 2018 Mar 13: 13-22. 2- Karimi P., Islami F., Anandasabapathy S., Freedman N.D., Kamangar F. Gastric cancer: descriptive epidemiology, risk factors, screening, and prevention. Cancer Epidemiol Biomarkers Prev. 2014;23(5):700-713. 3- Forman D., Burley V.J. Gastric cancer: global pattern of the disease and an overview of environmental risk factors. Best Pract Res ClinGastroenterol. 2006;20(4):633-649. 4- Ferlay J, Soerjomataram I, Ervik M, Dikshit R, Eser S, Mathers C, et al. GLOBOCAN 2012 v1.0, Cancer Incidence and Mortality Worldwide: IARC CancerBase No. 11. Lyon, France: International Agency for Research on Cancer; 2013. [Internet]. [cited 2014 Feb 22]. Available from: <http://globocan.iarc.fr/Pages/references.aspx>. 5- Ministry of Health and Population. Gharbiah Population Based Cancer Registry, Egypt. .Cancer in Egypt, triennial report of 2000-2002. 2007. MOH: Tanta, Egypt. 6-Alieldin N. NCI hospital-based registry 2002-2010 [Internet]. [cited 2014 Feb23].Availablefrom:<http://nci.cu.edu.eg/App_Files/registry/NCI_registry%202002-2010.pdf>. 7-Freedman L, Edwards B, Ries L, Young J, editors. Cancer incidence in four member countries (Cyprus, Egypt, Israel, and Jordan) of the Middle East Cancer Consortium (MECC) Compared with US SEER. National Cancer Institute, 2006. NIH Pub. No. 06-5873. Bethesda, MD [Internet]. [cited 2014 Feb 22]. 8- Zhou XM, Wong BC, Fan XM, Zhang HB, Lin MC, Kung HF, et al. Non-steroidal anti-inflammatory drugs induce apoptosis in gastric cancer cells through upregulation of bax and bak. Carcinogenesis. 2001;22:1393-97 9-Sasazuki S, Inoue M, Iwasaki M, Otani T, Yamamoto S, Ikeda S, et al. Effect of helicobacter pylori infection combined with cagA and pepsinogen status on gastric cancer development among Japanese men and women: A nested case-control study. Cancer Epidemiol. Biomarkers Prev. 2006;15:1341-47. 10- Tomonaga M, Oka M, Narasaki F, Fukuda M, Nakano R, Takatani H, et al. The multidrug resistance-associated protein gene confers drug resistance in human gastric and colon cancers. Jpn J Cancer Res. 1996;87:1263-70. 11-Buckland G, Travier N, Huerta JM, et al. Healthy lifestyle index and risk of gastric adenocarcinomaintheEPIC cohort study.IntJ Cancer. 2015;137(3):598-606. 12-Massarrat S, Stolte M. Development of gastric cancer and its prevention. Arch Iran Med. 2014;17(7):514-520. 13-Zhang ZX, ,Gu XZ, , Yin WB, , Huang GJ, , Zhang DW, , Zhang RG. Randomized clinical trial on the combination of preoperative irradiation and surgery in the treatment of adenocarcinoma of gastric cardia (AGC)-report on 370 patients. Int J RadiatOncolBiolPhys 1998; 42: 929-34. 14- Macdonald JS, , Smalley SR, , Benedetti J, , Hundahl SA, , Estes NC, , Stemmermann GN, et al. . Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med 2001; 345: 725-30. 15- M Fan W Hu Z Zhang. Chemoradiation for gastric cancer: controversies, updates and novel techniques. Br J Radiol July 2015; ( 88(1051).